CLINICAL TRIAL: NCT01821521
Title: A Randomized, Open Label, Single-dose, 2x2 Crossover Study to Investigate a Pharmacokinetics Between S-pantoprazole 20mg and Pantoprazole 40mg in Healthy Male Subjects
Brief Title: Investigate a Pharmacokinetics Between S-pantoprazole 20mg and Pantoprazole 40mg in Healthy Male Subjects
Acronym: S-Pantoprazole
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AGSPT_L20PK
Record Dates: First submitted 2013-03-25; First posted 2013-04-01 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AGSPT_L20 (Experimental): tablet, q.d.
  Interventions: Drug: AGSPT_L20
- Pantoloc 40mg (Active Comparator): tablet, q.d.
  Interventions: Drug: Pantoloc 40mg

INTERVENTIONS:
Drug: AGSPT_L20
  Arms: AGSPT_L20
Drug: Pantoloc 40mg
  Arms: Pantoloc 40mg

SUMMARY:
Primary object : Evaluate pharmacokinetic property administered S-pantoprazole 20mg and Pantoprazole 40mg in healthy male subjects

Secondary object : Evaluate safety administered S-pantoprazole 20mg and Pantoprazole 40mg in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy males 20 to 45 years at screening.
* BMI : 19kg/m2 ~ 26kg/m2
* Blood Pressure : "140 > sitting SBP ≥ 90mmHg, 90 > sitting DBP ≥ 60mmHg"

Exclusion Criteria:

* Have history of significant hepatic, renal, gastrointestinal, pulmonary, musculoskeletal, endocrine, neuropsychiatric, hematologic, cardiovascular diseases
* Have a gastrointestinal disease(ex : Crohn's disease, gastrointestinal ulcer)or surgery(except for Appendectomy, Hernia repair) affected the absorption of medications
* Have history of GERD, Gastric ulcer, Duodenal ulcer
* Hypersensitivity reactions to drugs or clinically significant hypersensitivity reactions in the history of benzimidazole(ex:pantoprazole, NSAID, antibiotic)
* Have a history of drug abuse
* Unusual diet affected the absorption, distribution, metabolism, excretion of medications
* Subject who treated with any investigational drugs within 90 days before the administration of investigational drug
* Subject who takes inhibitors and inducers of drug metabolizing enzyme (Barbiturates etc.) within 30days
* Previously donate whole blood within 60 days or component blood within 30 days or transfusion within 30 days
* Subject who have taken habitually caffeine (caffeine > 5 units/day)
* Subject who have drunken habitually (alcohol > 21 units/week, 1 unit = pure alcohol 10ml)or who are unable to quit drinking during this study or smoker
* Subjects deemed ineligible by investigator based on other reasons

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Cmax | 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24 hours
AUClast | 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24 hours

SECONDARY OUTCOMES:
AUCinf | 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24 hours
Tmax | 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24 hours
T1/2β | 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea